CLINICAL TRIAL: NCT03649217
Title: Active Limb Orthosis for Home-Use Stroke Hemiparetic Gait Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Moterum Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Moterum-iStride
Record Dates: First submitted 2018-08-06; First posted 2018-08-28 (Actual); Results first posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2020-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- wearing the iStride device (Experimental): The training will consist of four weeks of training with three training sessions performed each week. The training sessions will consist of up to thirty minutes of training with the iStride on, with breaks between walking sessions and as needed if the subject requests an additional break. Subjects will place the device on their foot in which they have the shortest step length, as measured during the pre-training gait analysis. This is typically the healthy side foot. There will also be several follow up visits following the final testing session.
  Interventions: Device: wearing the iStride device

INTERVENTIONS:
Device: wearing the iStride device — The device mimics the actions of the split-belt treadmill, but can be used during over-ground walking and in one's own home, thus enabling long-term training. This device does not require any external power and is completely passive; all necessary forces are redirected from the natural forces present during walking since it utilizes the wearer's weight to generate its movements. This research aims to test the iStride on individuals with stroke in their own home in order to determine if the related effects that we saw in the clinic, can also benefit patients at home.

SUMMARY:
The objective of this research is to test a passive shoe to correct gait in individuals with asymmetric walking patterns. This will be done in a clinic and within their own home. Individuals with central nervous system damage, such as stroke, often have irregular walking patterns and have difficulty walking correctly. Recent research has shown that using a split-belt treadmill can create after-effects that temporarily correct the inefficient walking patterns. However, the corrected walking pattern does not efficiently transfer from the treadmill to walking over ground. The iStride, formerly known as the Gait Enhancing Mobile Shoe (GEMS), may allow a patient to practice walking in many different locations, such as their own home, which we hypothesize will result in a more permanent transfer of learned gait patterns. To enable long-term use, our proposed shoe design is passive and uses the wearer's natural forces exerted while walking to generate the necessary motions.

DETAILED DESCRIPTION:
Hemiparesis and other impairments are a frequent and disabling consequence of stroke and can lead to asymmetric and inefficient walking patterns. Training on a split-belt treadmill, which has two separate treads driving each leg at a different speed, can correct gait asymmetries post-stroke. However, the effects of split-belt treadmill training only partially transfer to everyday walking over ground and extended training sessions are required to achieve long-lasting effects. Our previous studies suggest that the iStride device that has been developed in our laboratory can be used as an alternative gait training device for people with stroke. The iStride device mimics the actions of the split-belt treadmill, but can be used during over-ground walking and in one's own home, thus enabling long-term training. The iStride device does not require any external power and is completely passive; all necessary forces are redirected from the natural forces present during walking since it utilizes the wearer's weight to generate its movements. While the movements of the iStride device are similar to the split belt treadmill, and the iStride device generates a similar aftereffect, the efficacy of this shoe in modifying the gait of an individual with stroke is not yet verified. This research aims to continue to test the iStride device on individuals with stroke to determine if the related effects in a clinic setting, are also beneficial and safe in a home environment.

In this study, we will test the efficacy of the iStride device on individuals with stroke in the clinic and within their own home. Efficacy will be evaluated based on the change in gait coordination and also based on subjects' self-reported comfort on the device. We predict that the iStride device will result in changes to interlimb coordination of gait and prove to be a safe and effective device to be used in ones' home.

The asymmetric nature of hemiparetic gait can have a large impact on functional walking ability. For example, swing phase asymmetry is a significant predictor of hemiparetic walking performance because it strongly correlates with stages of motor recovery, walking speed, and falls. Another measure of temporal asymmetry - double support duration - is similarly correlated with walking speed. In addition, spatial (e.g. step length) asymmetry is associated with decreased propulsive force on the paretic leg, which limits forward motion of the body and reduces gait efficiency. The importance of gait efficiency should not be understated - the elevated energy demands of hemiparetic gait combined with physical deconditioning post-stroke can greatly limit performance of activities of daily living, contributing to poor cardiovascular fitness and metabolic syndrome. In turn, this can increase the risks of a second stroke or cardiovascular event and is associated with increased morbidity and mortality rates. Therefore, improving gait symmetry should be an important goal for therapy, to not only improve functional mobility and reduce injury, but also to enhance general health and well-being post-stroke.

Practicing walking on a split-belt treadmill can correct abnormal interlimb coordination of gait in individuals with hemiparesis following stroke or other central nervous system lesions. Asymmetric gait can manifest as a spatial asymmetry, in which steps taken on one side are longer than those on the other. It can also manifest as a temporal asymmetry, where the timing is uneven on the paretic and non-paretic sides. Temporal asymmetries are often measured as differences in the duration of double support periods, which are the amount of time both feet are simultaneously contacting the ground and are measured separately for the paretic and non-paretic sides. The iStride device is designed to cause changes in both spatial and temporal gait symmetry. We predict that the iStride device would cause the steps on the side with the iStride device to be larger since individuals would compensate for the backward rolling motion by placing their foot farther forward in stance, thus increasing the distance between the two feet. Similarly, since the stride is longer, it may also shorten the duration of stance relative to the other side. With shortened stance duration, the amount of time spent in double-support at the end of stance would likely decrease as well.

Although the original idea of the iStride device is derived from the motion of the split-belt-treadmill, there are distinct differences between walking on the device and walking on a split-belt treadmill with asymmetric belt velocities. While the body's velocity relative to ground is zero on a split-belt treadmill, the relative velocity of the iStride device is non-zero and forward. The device forces the wearer's foot forward or backward whereas the treadmill moves both feet backward, but at different speeds. For both the split-belt treadmill and the iStride device, the relative velocity between both feet is similar and the backward-moving iStride device takes the place of the faster tread.

We hypothesize that training over ground will lead to a change in the interlimb coordination in individuals with asymmetric gait and allow individuals to develop a more persistent symmetric gait. There are several differences between training on ground and a treadmill, such as visual flow and vestibular information signaling forward movement that likely limit the expression of learning in the over-ground context when trained on a treadmill. Visual cues appear to be particularly important for context awareness. Visual cues, coupled with prior experience, are so powerful that predictive postural responses cause an individual to stumble when stepping onto an escalator that is not moving. The body has learned an internal model that expects an acceleration when stepping onto an escalator, but when that acceleration does not occur, the person stumbles. A study of split-belt walking showed that transfer to over-ground walking is enhanced when subjects are blindfolded during training on the treadmill and tested over ground. Since blindfolding eliminates visual cues about the environment, this also suggests that vision is a key factor in determining the context-dependence of learning. Since it is not realistic to blindfold stroke patients during gait training, we designed the iStride device so that training could occur during over-ground walking, thus visual cues during training and later walking over ground would be the same.

Data from control subjects using an earlier version of the iStride device (referred to as GEMS at the time) has been published and a video of this previous version can be found at http://reedlab.eng.usf.edu/publications/handzic2011GEMS.mp4. In this study, we found that this earlier version of the device was capable of changing step length as predicted, however the previous design was too heavy and too tall to be considered practical for testing in stroke populations. The current version of the iStride device produces similar motion to the previous version, but it weighs less (under 1 kg) and is shorter (~4.4 cm). We will test the efficacy of wearing the current iStride device on gait coordination during walking over ground on individuals with stroke in the clinic and within their own home. All walking will be performed while subjects are closely guarded by an experienced physical therapist to prevent falling. The effects of the iStride device on gait coordination will be compared to those induced on a split-belt treadmill.

The proposed project represents one of the first attempts to build a device that corrects walking symmetry while walking over ground. Not only would this allow people to experience gait corrections while performing normal movements, but the simplicity and relative low cost of these devices would also open up potential opportunities to train at home (for high-functioning individuals with supervision) and in clinics where a split-belt treadmill is not available. The studies outlined here will establish whether the iStride device is capable of changing interlimb coordination of gait, and whether individuals with stroke can use these devices for rehabilitation purposes. This work will thus build the foundation for future training studies examining the effectiveness of long-term use of the iStride device for improving symmetric walking patterns.

The question that this study targets is the modification of human walking patterns for use in stroke rehabilitation. It is our ultimate objective to show that the iStride device can change a person's temporal and spatial gait asymmetry into a symmetric gait. We have demonstrated this in a clinic setting, and now we will test the device within the participants own home. Our points of reference are results obtained by previous studies with split-belt treadmills. We are also interested in how altering the interface between a foot and the ground influences the adaptation to new walking patterns.

ELIGIBILITY:
Inclusion Criteria:

* age 21-80
* one or more cerebral strokes, but all strokes on same side
* a stroke at least 6 months prior to enrollment
* Gait asymmetry, but able to walk independently with or without a cane
* Not currently receiving physical therapy
* no evidence of severe cognitive impairment that would interfere with understanding the instructions
* no evidence of one-sided neglect, affecting ambulation
* At least 25 feet of walking space in home (does not need to be a straight line)
* Weight does not exceed 250 lbs

Exclusion Criteria:

* uncontrolled seizures
* metal implants (stents, clips, pacemaker)
* pregnancy
* History of a neurological disorder other than stroke ( Parkinson's, MS)
* Chronic Obstructive Pulmonary Disease
* Uncontrolled blood pressure
* Head injury in the past 90 days
* A myocardial infarction within the last 180 days
* Cannot rely on a rolling walker for ambulation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Rashford, PT, Study Director — Moterum Technologies, LLC
Locations (4):
- United States (4):
  - University of South Florida, Tampa, Florida
  - homes throughout Charlotte, NC, Charlotte, North Carolina
  - homes throughout Memphis, TN, Memphis, Tennessee
  - homes throughout Burlington, VT, Burlington, Vermont

REFERENCES:
- [Background] Handzic I, Barno EM, Vasudevan EV, Reed KB. Design and Pilot Study of a Gait Enhancing Mobile Shoe. Paladyn. 2011 Dec 1;2(4):10.2478/s13230-012-0010-7. doi: 10.2478/s13230-012-0010-7. PMID 24371521
- [Background] Handzic I, Vasudevan E, Reed KB. Developing a Gait Enhancing Mobile Shoe to Alter Over-Ground Walking Coordination. IEEE Int Conf Robot Autom. 2012 May;2012:4124-4129. doi: 10.1109/ICRA.2012.6225346. PMID 23484067
- [Background] Kim S, Handzic I, Huizenga D, Edgeworth R, Lozinski M, Ramakrishnan T, & Reed KB,
- [Background] Handzic I, Reed KB. Comparison of the passive dynamics of walking on ground, tied-belt and split-belt treadmills, and via the Gait Enhancing Mobile Shoe (GEMS). IEEE Int Conf Rehabil Robot. 2013 Jun;2013:6650509. doi: 10.1109/ICORR.2013.6650509. PMID 24187324
- [Background] Kim SH, Huizenga DE, Handzic I, Ditwiler RE, Lazinski M, Ramakrishnan T, Bozeman A, Rose DZ, Reed KB. Relearning functional and symmetric walking after stroke using a wearable device: a feasibility study. J Neuroeng Rehabil. 2019 Aug 28;16(1):106. doi: 10.1186/s12984-019-0569-x. PMID 31455358
- [Derived] Darcy B, Rashford L, Tsai NT, Huizenga D, Reed KB, Bamberg SJM. One-year retention of gait speed improvement in stroke survivors after treatment with a wearable home-use gait device. Front Neurol. 2024 Jan 11;14:1089083. doi: 10.3389/fneur.2023.1089083. eCollection 2023. PMID 38274885
- See also: Additional information on a related stroke rehabilitation shoe. — http://reedlab.eng.usf.edu/iStrideDevice/
- See also: Commercial information about the iStride(TM) Device — https://moterum.com/relearn-to-walk/

RESULTS

PARTICIPANT FLOW:
Groups:
- Wearing the iStride Device: The training will consist of four weeks of training with three training sessions performed each week. The training sessions will consist of up to thirty minutes of training with the iStride on, with breaks between walking sessions and as needed if the subject requests an additional break. Subjects will place the device on their non-paretic foot. There will also be five follow up visits following the final testing session: one-week, one-month, three-months, six-months, and twelve-months
  Wearing the iStride device: The device mimics the actions of the split-belt treadmill, but can be used during over-ground walking and in one's own home, thus enabling long-term training. This device does not require any external power and is completely passive; all necessary forces are redirected from the natural forces present during walking since it utilizes the wearer's weight to generate its movements. This research aims to test the iStride on individuals with stroke in their own home in order to determine if the related effects that we saw in the clinic, can also benefit patients at home.
Period: Overall Study
Arm/Group | Wearing the iStride Device
Started | 23
Completed | 21
Not Completed | 2
Not completed — subject had severe ataxia not initially found | 1
Not completed — subject had cognitive issues not initially found | 1

BASELINE CHARACTERISTICS:
Arm/Group | Wearing the iStride Device
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.67 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Ten Minute Walk Test (10MWT)
Description: This test is to also help determine gait velocity/speed.
Time Frame: Difference between baseline assessment at start and one week post
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Arm/Group | Wearing the iStride Device
Number analyzed (Participants) | 21
meters per second (m/s) | 0.551 (0.245)
Statistical Analysis 1: Comparison: Wearing the iStride Device; Test type: Superiority; p = .0001, ANOVA

2. Primary Outcome: Change in Timed up and Go (TUG)
Description: This will provide a clinical assessment on gait speed/velocity. This also requires both static and dynamic balance as the participant will rise from a chair and sit down in a chair when the complete the test. The TUG test provides us different score assessments to help determine if a patient can, for example, cross a crosswalk safely.
Time Frame: Difference between baseline assessment at start and one week post
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Wearing the iStride Device
Number analyzed (Participants) | 21
seconds | 19.2 (8.06)
Statistical Analysis 1: Comparison: Wearing the iStride Device; Test type: Superiority; p = .0001, ANOVA

3. Secondary Outcome: Change in Berg Balance Scale
Description: This will provide a clinical assessment on balance using the total Berg Balance Scale. Scores range from 0 (least balance) to 56 (best balance).
Time Frame: Difference between baseline assessment at start and one week post
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Wearing the iStride Device
Number analyzed (Participants) | 21
scores on a scale | 43.52 (6.41)
Statistical Analysis 1: Comparison: Wearing the iStride Device; Test type: Superiority; p = .001, ANOVA

4. Secondary Outcome: Change in Functional Gait Assessment (FGA)
Description: The FGA measures both balance and walking ability with scores ranging from 0 (least ability) to 30 (highest ability).
Time Frame: Difference between baseline assessment at start and one week post
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Wearing the iStride Device
Number analyzed (Participants) | 21
scores on a scale | 15 (4.89)
Statistical Analysis 1: Comparison: Wearing the iStride Device; Test type: Superiority; p = .0002, ANOVA

5. Secondary Outcome: Change in Stroke Specific Quality of Life
Description: Stroke Specific Quality of Life will collect data on the psychosocial aspect of improvement to help look at the overall quality of life. The total score ranges from 49 to 245, with higher scores indicating a better quality of life.
Time Frame: Difference between baseline assessment at start and one week post
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Wearing the iStride Device
Number analyzed (Participants) | 21
scores on a scale | 165.05 (23.84)
Statistical Analysis 1: Comparison: Wearing the iStride Device; Test type: Superiority; p = .006, ANOVA

ADVERSE EVENTS:
Time Frame: six months
Arm/Group | Wearing the iStride Device
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wearing the iStride Device (N=21)
fall (Psychiatric disorders) | 1 (21) — The participant began to feel dizzy while walking and experienced a controlled fall into the chair. The participant was not injured. Of note, this participant had severe ataxia with vestibular symptoms in addition to stroke-related hemiparesis.
fall (Psychiatric disorders) | 1 (21) — The participant had a loss of balance that led to a controlled fall onto the floor. No injuries were sustained and, afterward, she was able to continue ambulating with the gait device for a total of 25 minutes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03649217/Prot_SAP_001.pdf